CLINICAL TRIAL: NCT01413945
Title: Evaluation of the Ileocecal Valve in Patients With and Without Irritable Bowel Syndrome.(IBS)
Brief Title: Ileocecal Sphincter Reflex by Cecal Distension During Colonoscopy
Status: Terminated | Type: Observational
Why Stopped: Not able to enroll enough patients in this study
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Larry Miller, Principal Investigator, Northwell Health
Other Study IDs: 13-216B
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: Ileocecal valve; Irritable bowel syndrome; small bowel bacteria
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal volunteers: Normal volunteers without Irritable bowel syndrome who are undergoing screening colonoscopy.
- Irritable bowel syndrome: Patients with Irritable bowel syndrome are undergoing colonoscopy as standard of care.

SUMMARY:
The aim of the current study is to test the hypothesis that patients with IBS may have a defective ICV pressures and may have small bowel bacterial overgrowth. The goal of the current study is to identify the role and competence of ileocecal valve (ICV) in patients with irritable bowel syndrome.

The primary objective is to measure the pressure of the ileocecal valve in patients with and without irritable bowel syndrome (IBS). The Ileocecal valve reflux pressures during air insufflation of cecum will be used.

DETAILED DESCRIPTION:
This is an outpatient study. There will be no requirement to stay overnight in the hospital. The research will be conducted in the gastroenterology section of the department of Medicine in North shore university hospital and in North shore long island Jewish medical center. Both these hospitals are tertiary care centers with adequate facilities for the safe and appropriate conduct of this research. Participants must meet all eligibility criteria and sign the consent form before enrolling in the study. This is a cohort study with 2 groups (patients with IBS and participants without IBS). Patients will be enrolled into one of these two categories based on their medical history, signs and symptoms and questionnaire. There are no controlled compounds used in this study. There is no treatment involved in this study. There are 2 study related visits per subject.

Based on questionnaire we plan to recruit 25 participants who meet the criteria of IBS and 25 participants who do not meet the criteria of IBS (Total of 50 participants in the study). Patients with IBS are those who meet the criteria of IBS based on their symptoms and the responses to a validated ROME III - questionnaire. All other participants who do not meet the criteria for IBS are classified as non-IBS participants. All the participants should be having a clinically indicated colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of small bowel bacterial overgrowth or irritable bowel syndrome and who are undergoing routine colonoscopies or subjects who are undergoing routine colonoscopy and test positive for small bowel bacterial overgrowth will be candidates. If the patient has prior lactulose breath test done for clinical purposes then repeat lactulose breath test will not be required. If no prior lactulose breath test has been performed then it will be done as part of this research study. In addition patients who test negative for SBBO will be candidates for the control population.

Exclusion Criteria:

* Medications-Subjects on any medication that could affect the ileocecal valve high-pressure zone will be excluded; this includes use of prokinetic agents, current use of any antibiotics and anticholinergics. Patients will be excluded if the lactulose breath test is done on antibiotics or during the colonoscopy preparation.

GI symptoms, conditions and disorders: In addition exclusion criteria will include a history of ileocecal resection or disease affecting the colon and/or small bowel including crohn's disease, ulcerative colitis or diseases causing diarrhea.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with who are undergoing routine screening colonoscopies.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-06-21 (Actual); Primary Completion 2015-08-05 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Pressure generated in ICV during Cecal distention | 10-15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Larry S Miller, MD, Principal Investigator — Northwell Health
Locations (1):
- LIJ Medical Center- NSLIJ Health System, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GAZET RJ, JARRETT J. THE ILEOCAECO-COLIC SPHINCTER. STUDIES IN VITRO IN MAN, MONKEY, CAT, AND DOG. Br J Surg. 1964 May;51:368-70. doi: 10.1002/bjs.1800510519. No abstract available. PMID 14153394
- [Background] SINGLETON AO Jr, REDMOND DC 2nd, MCMURRAY JE. ILEOCECAL RESECTION AND SMALL BOWEL TRANSIT AND ABSORPTION. Ann Surg. 1964 May;159(5):690-4. doi: 10.1097/00000658-196405000-00006. No abstract available. PMID 14158913
- [Background] Jarrett RJ, Gazet JC. Studies in vivo of the ileocaeco-colic sphincter in the cat and dog. Gut. 1966 Jun;7(3):271-5. doi: 10.1136/gut.7.3.271. No abstract available. PMID 18668804
- [Background] Kelley ML Jr, Gordon EA, Deweese JA. Pressure responses of canine ileocolonic junctional zone to intestinal distention. Am J Physiol. 1966 Sep;211(3):614-8. doi: 10.1152/ajplegacy.1966.211.3.614. No abstract available. PMID 5927889
- [Background] Cohen S, Harris LD, Levitan R. Manometric characteristics of the human ileocecal junctional zone. Gastroenterology. 1968 Jan;54(1):72-5. No abstract available. PMID 5635439
- [Background] Castell DO, Cohen S, Harris LD. Response of human ileocecal sphincter to gastrin. Am J Physiol. 1970 Sep;219(3):712-5. doi: 10.1152/ajplegacy.1970.219.3.712. No abstract available. PMID 5450876
- [Background] Griffen WO Jr, Richardson JD, Medley ES. Prevention of small bowel contamination by ileocecal valve. South Med J. 1971 Sep;64(9):1056-8. doi: 10.1097/00007611-197109000-00006. No abstract available. PMID 5096285
- [Background] Pahlin PE, Kewenter J. Sympathetic nervous control of cat ileocecal sphincter. Am J Physiol. 1976 Aug;231(2):296-305. doi: 10.1152/ajplegacy.1976.231.2.296. PMID 961880
- [Background] Stremmel W, Kurpreugsch K, Langewitz W. [Hormonal and pharmacological modification of the ileocecal sphincter]. Chir Forum Exp Klin Forsch. 1977 Apr:45-8. German. PMID 618312
- [Background] King CE, Toskes PP. Small intestine bacterial overgrowth. Gastroenterology. 1979 May;76(5 Pt 1):1035-55. No abstract available. PMID 437407
- [Background] Rubin MR, Fournet J, Snape WJ Jr, Cohen S. Adrenergic regulation of ileocecal sphincter function in the cat. Gastroenterology. 1980 Jan;78(1):15-21. No abstract available. PMID 7350021